CLINICAL TRIAL: NCT02578121
Title: A Phase II Trial of a Novel Proteasome/IMiD Combination, Ixazomib, Pomalidomide, and Dexamethasone in Relapsed Multiple Myeloma Patients
Brief Title: UARK 2015-03 A Phase II Trial of a Novel Proteasome/IMiD Combination
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Investigator decided to close study without enrollment
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0203974
Record Dates: First submitted 2015-10-14; First posted 2015-10-16 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2017-01

CONDITIONS: Multiple Myeloma
Keywords: Relapsed; Response Rate; Progression free
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — ixazomib; pomalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ixazomib, Pomalidomide, Dexamethasone (Experimental): Protasome/IMiD combination of Ixazomib 4mg days 1, 8, and 15, Pomalidomide 4mg days 1-21 amd Dexamethasone 20 mg days 1, 8, 15 and 22 of a 28 day cycle
  Interventions: Drug: Ixazomib; Drug: Pomalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Ixazomib — 4.0 mg will be given on days 1, 8 and 15 of a 28 day cycle
Drug: Pomalidomide — 4.0 mg will be given on days 1-21 of a 28 day cycle
Drug: Dexamethasone — 20 mg will be given on days 1, 8, 15 and 22 of a 28 day cycle

SUMMARY:
The purpose of this study is to determine the efficacy of Ixazomib when combined with Pomalidomide and Dexamethasone, in terms of overall response rate in subjects with relapsed Multiple Myeloma

DETAILED DESCRIPTION:
This single arm, Phase II study will examine the efficacy and safety of the novel Proteasome/IMiD combination of Ixazomib 4mg days 1, 8, 15, Pomalidomide 4 mg days 1-21, Dexamethasone 20 mg days 1, 8, 15, and 22 of a 28 day cycle, in relapse patients. The long term aim being to develop a backbone regimen to which future novel targeted treatments may be added as part of a personalized medicine approach.

ELIGIBILITY:
Inclusion Criteria:

* Each patient must meet all of the following inclusion criteria to be enrolled in the study:

  * Male or female patients 18 years or older.
  * Voluntary written consent must be given before performance of any study related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.
  * Female patients who:

Are postmenopausal for at least 1 year before the screening visit, OR Are surgically sterile, OR If they are of childbearing potential, agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent form through 90 days after the last dose of study drug, AND Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [eg, calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception.)

* Male patients, even if surgically sterilized (ie, status post-vasectomy), must agree to one of the following: Agree to practice effective barrier contraception during the entire study treatment period and through 90 days after the last dose of study drug, OR Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence (eg, calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception.)
* Patients must have a diagnosis of relapsed and/or refractory multiple myeloma and must have received at least one line of prior therapy. Patients must be at least 14 days beyond the last multiple myeloma therapy and have recovered from acute toxicities of prior therapies measured by CTCAE (Version 4.0)
* Patients must have life expectancy of at least 3 months.
* Eastern Cooperative Oncology Group (ECOG) performance status and/or other performance status 0, 1, or 2.
* Patients must meet the following clinical laboratory criteria:

Absolute neutrophil count (ANC) > 1,000/mm3 and platelet count> 50,000/mm3. Platelet transfusions to help patients meet eligibility criteria are not allowed within 3 days before study enrollment. Total bilirubin <1.5 x the upper limit of the normal range (ULN). Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 3 x ULN. Calculated creatinine clearance > 30 mL/min (see APPENDIX C for the Cockcroft-Gault Equation).,

Exclusion Criteria:

- Patients meeting any of the following exclusion criteria are not to be enrolled in the study:

* Female patients who are lactating or have a positive serum pregnancy test during the screening period.
* Failure to have fully recovered (ie, < Grade 1 toxicity) from the reversible effects of prior chemotherapy.
* Major surgery within 14 days before enrollment.
* Radiotherapy within 14 days before enrollment. If the involved field is small, 7 days will be considered a sufficient interval.
* Central nervous system involvement.
* Infection requiring systemic antibiotic therapy or other serious infection within 14 days before study enrollment.
* Evidence of current uncontrolled cardiovascular conditions, including uncontrolled hypertension, uncontrolled cardiac arrhythmias, symptomatic congestive heart failure, unstable angina, or myocardial infarction within the past 6 months.
* Ongoing or active systemic infection, active hepatitis B or C virus infection, or known human immunodeficiency virus (HIV) positive.
* Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol.
* Known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent.
* Known GI disease or GI procedure that could interfere with the oral absorption or tolerance of oral medications including difficulty swallowing.
* Diagnosed or treated for another malignancy within 2 years before study enrollment or previously diagnosed with another malignancy and have any evidence of residual disease. Patients with non-melanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.
* Patient has > Grade 3 peripheral neuropathy, or Grade 2 with pain on clinical examination during the screening period.
* Participation in other clinical trials, including those with other investigational agents not included in this trial, within 21 days of the start of this trial and throughout the duration of this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-12; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Response rate after combination of Ixazomib, Pomalidomide and Dexamethasone therapy | 28 days
  Response rate will be assessed at baseline, with each scheduled study visit , including the exit visit.

CONTACTS AND LOCATIONS:
Overall Officials: Faith Davies, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Science, Little Rock, Arkansas, United States